CLINICAL TRIAL: NCT04603937
Title: A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared With Intravitreal Aflibercept in Participants With Visual Impairment Secondary to Treatment-naïve Diabetic Macular Edema (DME)
Brief Title: A Study to Evaluate the Efficacy, Durability, and Safety of KSI-301 Compared to Aflibercept in Participants With Diabetic Macular Edema (DME)
Acronym: GLIMMER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet primary endpoint
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P105; 2020-001063-82 (EudraCT Number)
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Kodiak; Vascular endothelial growth factor; Anti-VEGF; VEGF; Antibody biopolymer conjugate; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, low; Aflibercept; Eylea; Diabetes mellitus; Diabetes; Diabetic retinopathy; Diabetic macular edema; Macular edema; KSI-301
MeSH Terms: conditions — Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low; Diabetes Mellitus; Diabetic Retinopathy; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two treatment arms: KSI-301 or aflibercept.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For masking purposes, sham injections will be administered at every monthly visit if an active treatment is not administered. To preserve masking, two investigators are required for this study. The masked Investigator will be responsible for the examinations and safety assessments. The unmasked Investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 (Arm A) (Experimental): Intravitreal injection of KSI-301 (5 mg) once every 4 weeks for 3 monthly doses followed by an individualized dosing regimen (every 8 to 24 weeks) via intravitreal injection from Week 16 to Week 100.
  Interventions: Drug: KSI-301; Other: Sham Procedure
- Aflibercept (Arm B) (Active Comparator): Intravitreal injection of aflibercept (2 mg) once every 4 weeks for 5 monthly doses followed by aflibercept (2 mg) once every 8 weeks via intravitreal injection from Week 24 to 100.
  Interventions: Drug: Aflibercept; Other: Sham Procedure

INTERVENTIONS:
Drug: KSI-301 — Intravitreal Injection
  Arms: KSI-301 (Arm A)
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept (Arm B)
Other: Sham Procedure — The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This Phase 3 study will evaluate the efficacy, durability, and safety of KSI-301 compared to aflibercept in participants with treatment-naïve DME.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, double-masked, two-arm, multi-center non-inferiority study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in participants with treatment-naïve DME.

The primary endpoint will be assessed at Year 1; additional secondary endpoints for efficacy will be assessed at Years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Treatment-naïve diabetic macular edema, with vision loss and center involvement (if present) diagnosed within 9 months of screening.
3. BCVA ETDRS letter score between 78 and 25 (-20/25 to 20/320 Snellen equivalent), inclusive, in the Study Eye.
4. CST of ≥ 320 microns on SD-OCT (Heidelberg Spectralis or equivalent on other OCT instruments) as determined by the Reading Center.
5. Decrease in vision determined by the Investigator to be primarily the result of DME.
6. Type 1 or Type 2 diabetes mellitus and a HbA1c of ≤12%.
7. Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

1. Macular edema in the Study Eye considered to be secondary to a cause other than DME.
2. Active iris or angle neovascularization or neovascular glaucoma in the Study Eye.
3. High-risk proliferative diabetic retinopathy characteristics in the Study Eye.
4. History of Pan-retinal Photocoagulation (PRP) laser in the Study Eye within 3 months of screening.
5. Tractional retinal detachment in the Study Eye.
6. Active retinal disease other than the condition under investigation in the Study Eye.
7. Any history or evidence of a concurrent ocular condition present, that in the opinion of the Investigator could require either medical or surgical intervention or affect macular edema or alter visual acuity during the study (e.g., vitreomacular traction, epiretinal membrane).
8. Active or suspected ocular or periocular infection or inflammation in either eye at Day 1.
9. Any prior use of an approved or investigational treatment for DME in the Study Eye (e.g., anti-VEGF, intraocular or periocular steroids, macular laser photocoagulation).
10. Women who are pregnant or lactating or intending to become pregnant during the study.
11. Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg or diastolic value ≥100 mmHg while at rest.
12. Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
13. History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
14. Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (72):
- United States (40):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Vitreous Associates, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Retina Group of New England, Waterford, Connecticut
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, P.C., Marietta, Georgia
  - Retina Consultants of Hawaii, Inc, ‘Aiea, Hawaii
  - Retina Specialists of Idaho, Boise, Idaho
  - Talley Eye, Evansville, Indiana
  - Maine Eye Center, Portland, Maine
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Vitreoretinal Surgery PA, Minneapolis, Minnesota
  - Retina Consultants of NV, Henderson, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Vitreo Retinal Consultants, Hauppauge, New York
  - Retina-Vitreous Surgeons of Central NY, Liverpool, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Retina Associates of Western NY, Rochester, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - Cleveland Clinic Foundation, Cole Eye Institute, Cleveland, Ohio
  - Retina Consultants, LLC, Salem, Oregon
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Houston-(Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates (Round Rock), Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Houston - (Woodlands), The Woodlands, Texas
  - Retina Institute of Virginia, Richmond, Virginia
- Czechia (3):
  - OFTEX s.r.o., Pardubice
  - Vseobecna Fakultni, Prague
  - Lekarna BENU, Prague
- France (6):
  - CHRU Dijon Complexe Du Bocage, Dijon, Côte-d'Or
  - Hôpital de La Croix Rousse, Lyon, Rhône
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Paradis Monticelli, Marseille
  - Hôpital Lariboisière - Service Pharmacie , Essais cliniques - Aude Jacob, Paris
  - Fondation Rothschild, Paris
- Hungary (4):
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz , Josa Andras Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associates Kft, Budapest
- Israel (9):
  - Bnai Zion, Haifa
  - Rambam MC, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir MC, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan MC, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta HaShalom, Tel Aviv
  - Shamir Medical Center Assaf Harofeh, Tzrifin
- Italy (3):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Naples
- Poland (6):
  - Optimum Profesorskie Centrum Okulistyki, Gdansk, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne Im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowi, Katowice, Silesian Voivodeship
  - Oftalmika Sp. z o.o., Bydgoszcz
  - Dr Nowosielska Okulistyka i Chirurgia Oka, Warsaw
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Wałbrzych
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Emanuelli Research & Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 75 medical centers between September 2020 and January 2022. The first participant was enrolled on 30 September 2020 and the last on 31 January 2022.
Pre-assignment Details: Of 689 screened participants, 459 met eligibility criteria and were randomized to treatment. Two randomized subjects in KSI-301 arm never received treatment, so do not have reason for not completing treatment. Each participant contributed only one study eye to this study.
Period: Overall Study
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Started | 229 (The number of participants who started in KSI-301 (Arm A) reflects those who actually received the treatment.) | 228
Completed (Completed is defined as participants who completed treatment through Week 64.) | 208 | 204
Not Completed | 21 | 24
Not completed — Adverse Event | 9 | 10
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 5 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Subject did not meet inclusion criteria 1 so was withdrawn from the study | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set defined as all randomized subjects who received any study treatment (KSI-301 or aflibercept). Subjects will be analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B) | Total
Number analyzed (Participants) | 229 | 228 | 457
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 137 | 270
  >=65 years | 96 | 91 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.34) | 61.6 (9.90) | 61.9 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 79 | 176
  Male | 132 | 149 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 58 | 100
  Not Hispanic or Latino | 182 | 161 | 343
  Unknown or Not Reported | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 12 | 34
  White | 194 | 201 | 395
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 8 | 11 | 19
Geographic Region [Count of Participants; unit: Participants]
  North America | 149 | 147 | 296
  Rest of World | 80 | 81 | 161
BCVA in the Study Eye, Letters [Mean (Standard Deviation); unit: Letters] | 64.2 (11.43) | 64.3 (11.21) | 64.2 (11.31)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in BCVA
Description: Mean change in best-corrected visual acuity (BCVA) from baseline to the average of Weeks 60 and 64 (using Early Treatment Diabetic Retinopathy Study (ETDRS) Letters). Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Day 1 to Week 64
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 229 | 228
ETDRS Letters | 6.7 (0.80) | 11.5 (0.81)
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable true difference between KSI-301 and aflibercept participants to be considered non-inferior is 4.5 ETDRS letters, i.e. the non-inferiority margin; p > 0.9999, Mixed Models Analysis; MMRM model with treatment, visit, treatment by visit interaction, randomization stratification factors, and continuous baseline BCVA and OCT CST; Adjusted mean difference = -4.7, 95.04% CI 2-sided [-6.65 to -2.81], Standard Error of Mean 0.97

2. Secondary Outcome: Percentage of Patients With a ≥ 2-step Worsening on the ETDRS DRSS in Studies KS301P104 and KS301P105 Combined
Description: Percentage of patients with a ≥ 2-step worsening on the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 52 using last observation carried forward (LOCF) in Studies KS301P104 and KS301P105 combined. The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 52
Population: All randomized subjects in Studies KS301P104 and KS301P105 who received any study treatment (KSI-301 or aflibercept) with evaluable results at baseline and evaluable results on or prior to Week 52. The population for studies KS301P104 and KS301P105 are identical in terms of treatment indication and inclusion/exclusion criteria. Please refer to NCT04611152 to review demographics, other study details and adverse events for participants in KS301P104 study.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 433 | 437
Participants | 6 | 3
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable non-inferiority margin between KSI-301 and aflibercept subjects is 10% to be considered non-inferior, i.e. the non-inferiority margin is 10%; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haentzel test stratified by study identifier and randomization stratification variables; Difference of weighted percentages = 0.6, 95.04% CI 2-sided [-0.7 to 2] — Weighted percentages are based on weighted average of observed estimates across strata using CMH weights. The CI are based on the normal approximation to the binomial proportions

3. Secondary Outcome: Percentage of Patients With a ≥ 2-step Worsening on the ETDRS DRSS in Study KS301P105
Description: Percentage of patients with a ≥ 2-step worsening on the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 52 using last observation carried forward (LOCF) in Study KS301P105. The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 52
Population: All randomized subjects who received any study treatment (KSI-301 or aflibercept) with evaluable results at baseline and evaluable results on or prior to Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 218 | 218
Participants | 6 | 3
Statistical Analysis 1: Comparison: KSI-301 (Arm A) vs Aflibercept (Arm B); Test type: Non-Inferiority — The maximum clinically acceptable non-inferiority margin between KSI-301 and aflibercept subjects is 10% to be considered non-inferior, i.e the non-inferiority margin is 10%; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haentzel test stratified by randomization stratification variables; Difference of weighted percentages = 1.2, 95.04% CI 2-sided [-1.4 to 3.9] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Patients in the KSI-301 Arm on a Q8W, Q12W, Q16W, Q20W, or Q24W Treatment Interval
Description: Percentage of patients in the KSI-301 arm on a Q8W, Q12W, Q16W, Q20W, or Q24W treatment interval at the primary endpoint. Analyses include KSI-301 patients who completed a treatment interval from Week 56 onwards.
Time Frame: Week 56
Population: Analyses include KSI-301 patients who completed a treatment interval from Week 56 onwards.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Arm A)
Number analyzed (Participants) | 210
Participants
  Number of participants on the KSI-301 Q8W | 54
  Number of participants on the KSI-301 Q12W | 23
  Number of participants on the KSI-301 Q16W | 14
  Number of participants on the KSI-301 Q20W | 10
  Number of participants on the KSI-301 Q24W | 109

5. Secondary Outcome: Mean Number of Intravitreal Injections
Description: Mean number of intravitreal injections from Day 1 to Week 60
Time Frame: Day 1 to Week 60
Population: Safety Analysis Set includes all patients who received any study treatment (KSI-301 or aflibercept).
  Patients will be analyzed according to the study treatment they actually received. One patient was randomized to KSI-301, but received aflibercept.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 228 | 229
injections | 5.8 (1.64) | 9.2 (1.91)

6. Secondary Outcome: Mean Change in OCT CST
Description: Mean change in Optical Coherence Tomography (OCT) central subfield retinal thickness (CST) baseline to the average of Weeks 60 and 64
Time Frame: Day 1 to Week 64
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
Number analyzed (Participants) | 229 | 228
Microns | -154.7 (128.03) | -194.2 (154.44)

ADVERSE EVENTS:
Time Frame: Time Frame Adverse Events (AEs) reported through Week 64 or Early Termination (ET) if occurred before Week 64.
Description: One subject randomized to KSI-301 treatment arm received incorrect treatment of Aflibercept, so was included in the Aflibercept treatment arm for safety analyses. Therefore, for adverse event reporting, there are 228 subjects in KSI-301 treatment arm and 229 subjects in Aflibercept treatment arm.
Arm/Group | KSI-301 (Arm A) | Aflibercept (Arm B)
All-Cause Mortality (participants affected / at risk) | 4/228 | 6/229
Serious Adverse Events (participants affected / at risk) | 53/228 | 57/229
Other Adverse Events (participants affected / at risk) | 113/228 | 104/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=228) | Aflibercept (Arm B) (N=229)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (4) | 4 (4)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 4 (5)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract - Study Eye (Eye disorders) | 1 (1) | 1 (1)
Angle closure glaucoma - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)
Cataract - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis - Fellow Eye (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage - Fellow Eye (Eye disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (2)
Death (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
Osteomyelitis (Infections and infestations) | 3 (3) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Localised infection (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis - Fellow Eye (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (3)
Endophthalmitis - Study Eye (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
West Nile viral infection (Infections and infestations) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalomalacia (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Arm A) (N=228) | Aflibercept (Arm B) (N=229)
Cataract - Study Eye (Eye disorders) | 33 (34) | 15 (15)
Conjunctival haemorrhage - Study Eye (Eye disorders) | 22 (25) | 8 (10)
Diabetic retinal oedema - Fellow Eye (Eye disorders) | 14 (16) | 24 (25)
Cataract - Fellow Eye (Eye disorders) | 12 (12) | 12 (12)
Diabetic retinal oedema - Study Eye (Eye disorders) | 12 (15) | 4 (5)
COVID-19 (Infections and infestations) | 32 (33) | 34 (34)
Diabetes mellitus (Metabolism and nutrition disorders) | 22 (23) | 22 (23)
Hypertension (Vascular disorders) | 23 (24) | 23 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04603937/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT04603937/SAP_001.pdf